CLINICAL TRIAL: NCT06568302
Title: A Global Open-label Extension Study to Observe the Long-term Safety and Efficacy of SerpinPC in Subjects with Hemophilia Who Completed a Sponsored SerpinPC Clinical Trial
Brief Title: The Long-term Safety and Efficacy of SerpinPC in Subjects with Hemophilia Who Completed a Sponsored SerpinPC Clinical Trial
Acronym: PRESent-6
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated due to business and strategic decision.
Sponsor: ApcinteX Ltd (Industry)
Collaborators: Centessa Pharmaceuticals plc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AP-0106; 2023-509965-19 (Other: EU CT Number)
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Hemophilia a; Hemophilia B; Hemophilia a with Inhibitor; Hemophilia B with Inhibitor
Keywords: Hemophilia; SerpinPC
MeSH Terms: conditions — Hemophilia A; Hemophilia B | interventions — Protein C

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- SerpinPC (Experimental): Participants will receive SerpinPC 1.2 milligrams/kilograms (mg/kg) subcutaneous injection every 2 weeks (Q2W) once they have completed treatment in a SerpinPC parent study.
  Interventions: Drug: SerpinPC

INTERVENTIONS:
Drug: SerpinPC — Administered as SC injection.
  Other Names: Activated Protein C (APC) inhibitor

SUMMARY:
The purpose of the study is to evaluate the efficacy, safety, tolerability and pharmacokinetic (PK) profile of prophylactic SerpinPC in participants with hemophilia

ELIGIBILITY:
Inclusion Criteria:

* Male participants greater than or equal to (>=) 12 and less than or equal to (<=) 65 years of age at the time of informed consent
* Completed participation in a sponsored SerpinPC hemophilia clinical trial and, in the opinion of the investigator, was compliant with the study including compliance with diary entries.
* Capable of providing written informed consent (adolescent assent and parent/guardian consent when appropriate) for participation

Exclusion Criteria:

* Previous deep vein thrombosis and pulmonary embolism, myocardial infarction, or embolic stroke
* Participation in another interventional clinical trial, except for SerpinPC trials
* Any other significant conditions or comorbidities that, in the opinion of the investigator, would make the subject unsuitable for enrolment or could interfere with participation in or completion of the study
* Treatment with anticoagulant or antiplatelet drugs

Ages: 12 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2024-07-11 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2025-01-29 (Actual)

PRIMARY OUTCOMES:
Treated bleeds, expressed as annualized bleeding rate (ABR) | Month 0 to Month 25 or Early termination

SECONDARY OUTCOMES:
Treated spontaneous bleeds (expressed as ABR) | Month 0 to Month 25 or Early termination
Treated spontaneous joint bleeds (expressed as ABR) | Month 0 to Month 25 or Early termination
All bleeds requiring treatment (expressed as ABR, ie, all treated bleeds and all bleeds that would ordinarily be treated with factor concentrate/bypass agent if therapy were available) | Month 0 to Month 25 or Early termination
Total coagulation factor and/or bypass product consumption | Month 0 to Month 25 or Early termination

CONTACTS AND LOCATIONS:
Locations (2):
- ARENSIA Exploratory Medicine LLC, Tbilisi, Georgia
- Institute of Oncology, ARENSIA Exploratory Medicine, Chisinau, Moldova

IPD SHARING:
Plan to Share IPD: No